CLINICAL TRIAL: NCT06541808
Title: Balance, Sensory Modulation, and Autonomic Response to Different Dosages of Non-invasive Mechanical Vagal Stimulation in Healthy Adults
Brief Title: Balance, Autonomic Response, and Sensory Modulation to Dosage of Mechanical Vagal Stimulation in Healthy Adults
Acronym: BARVANS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Giacomo Carta, Postdoc PhD Researcher, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK Nr: 1349/2024
Record Dates: First submitted 2024-07-03; First posted 2024-08-07 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Vagus Nerve Autonomic Disorder; Heart Rate; Pain; Equilibrium; Disorder, Labyrinth; Microbial Colonization
Keywords: Non-invasive Vagus Nerve stimulation; Heart Rate; Equilibrium; Pain modulation; Gut microbiota
MeSH Terms: conditions — Pain; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mechanical Vagus Nerve Stimulation (Low Intensity) (Experimental): 4 minutes of mechanical vagal stimulation (2 minutes on each side) administered only once along the entire experiment
  Interventions: Other: mechanical Vagus Nerve Stimulation (Low Intensity)
- mechanical Vagus Nerve Stimulation (Intermediate Intensity) (Experimental): 12 minutes of mechanical vagal stimulation(3 sessions of 2 minutes of stimulation, with 2 minutes of rest for each side) administered only once along the entire experiment
  Interventions: Other: mechanical Vagus Nerve Stimulation (Intermediate Intensity)
- mechanical Vagus Nerve Stimulation (High Intensity) (Experimental): 16 minutes of mechanical vagal stimulation (8 minutes on each side) administered only once along the entire experiment
  Interventions: Other: mechanical Vagus Nerve Stimulation (High Intensity)
- Sham Vagus Nerve Stimulation (Sham Comparator): Participants will be treated with a fake vagus stimulation not able to stretch the vagus nerve
  Interventions: Other: Sham mechanical Vagus Nerve Stimulation

INTERVENTIONS:
Other: mechanical Vagus Nerve Stimulation (Low Intensity) — The stimulation consists of a combination of normal neck movements, performed in a comfortable supine position, which can selectively stimulate the VN. In particular. The participant will be stimulated supine on a comfortable massage/treatment bed with the experimenter standing at the cranial short side of the bed. All the neck movements will be gently performed with a combination of upper cervical flexion and contralateral lateral flexion to load the intracranial portion of the vagus nerve. The ipsilateral neck rotation will be combined to load the cervical tract of the nerve. Keeping the participant's head in the final movements combination the upper abdomen will be gently moved caudally to load the thoracic tract and intermittent gentle impulses 1 each second will be administered. The stimulation will be provided for 2 consecutive minutes for each side, only once for the experiment duration.
  Arms: mechanical Vagus Nerve Stimulation (Low Intensity)
Other: mechanical Vagus Nerve Stimulation (Intermediate Intensity) — The stimulation consists of a combination of normal neck movements, performed in a comfortable supine position, which can selectively stimulate the VN. In particular. The participant will be stimulated supine on a comfortable massage/treatment bed with the experimenter standing at the cranial short side of the bed. All the neck movements will be gently performed with a combination of upper cervical flexion and contralateral lateral flexion to load the intracranial portion of the vagus nerve. The ipsilateral neck rotation will be combined to load the cervical tract of the nerve. Keeping the participant's head in the final movements combination the upper abdomen will be gently moved caudally to load the thoracic tract and intermittent gentle impulses 1 each second will be administered. The stimulation will be provided for 3 sessions of 2 minutes, with 2 minutes of rest for each side. stimulation will be provided only once for the experiment duration.
  Arms: mechanical Vagus Nerve Stimulation (Intermediate Intensity)
Other: mechanical Vagus Nerve Stimulation (High Intensity) — The stimulation consists of a combination of normal neck movements, performed in a comfortable supine position, which can selectively stimulate the VN. In particular. The participant will be stimulated supine on a comfortable massage/treatment bed with the experimenter standing at the cranial short side of the bed. All the neck movements will be gently performed with a combination of upper cervical flexion and contralateral lateral flexion to load the intracranial portion of the vagus nerve. The ipsilateral neck rotation will be combined to load the cervical tract of the nerve. Keeping the participant's head in the final movements combination the upper abdomen will be gently moved caudally to load the thoracic tract and intermittent gentle impulses 1 each second will be administered. The stimulation will be provided for 8 consecutive minutes for each side, only once for the experiment duration.
  Arms: mechanical Vagus Nerve Stimulation (High Intensity)
Other: Sham mechanical Vagus Nerve Stimulation — Participants will be treated with a fake vagus stimulation by letting the operator hold the neck of the participant in one hand and placing the other hand on the abdomen without any stretch on the vagus nerve
  Arms: Sham Vagus Nerve Stimulation

SUMMARY:
The vagus nerve (VN) plays a crucial role in regulating vital functions (heart rate, blood pressure, digestion, and immune response) and maintaining communication between internal organs and the brain. Recent studies have highlighted the therapeutic potential of VN stimulation (VNS) in treating various conditions such as drug-resistant epilepsy, postural control deficit, COVID-19 infection, chronic pain, and intestinal disorders. In addition, there is growing evidence that the molecules released by the VN neurons affect the function of the gut microbiota and that the molecules released by the bacteria in our gut affect the activity of the VN neurons. In particular, Dr. Giacomo Carta (the leader of this study) has shown how painless neck movements, i.e. mechanical VNS (mVNS), can be applied without adverse effects, representing a potential alternative to invasive methods commonly used today. To further investigate the impact of this novel mVNS, this study aims to evaluate the changes induced by three mVNS protocols on physiological parameters such as resting heart rate, and Heart Rate Variability (HRV) at rest, balance in standing, the perceived intensity of mechanical stimuli using the established clinical method of QST (quantitative sensory testing), fecal transit speed, and the molecular composition of stool (for this, stool samples are analyzed). In particular, stool analysis is very relevant for understanding normal digestion. The present research aims to define the optimal intensity of mVNS and to investigate the therapeutic potential of VNS in the treatment of autonomic dysfunction (such as too low or too high heart rate, too low or too fast digestion, throbbing headaches), as well as falls prevention and pain.

DETAILED DESCRIPTION:
mechanical VNs in humans, induced by a combination of non-painful physiological neck movements, effectively reduces the HR at rest in humans, without any side effects in the short- and long-term. Indeed, HR reduction is a proxy for the VN increased activity among healthy subjects and patients with systemic diseases or autonomic diseases. Mechanical VNs had been successfully adopted in two clinical trials among chronic pain patients (NCT05345496, NCT05360589), but due to the early stage of these new VNs and the clear advantages of this method, studies refining the stimulation protocol are suitable. Thus, the study aims to investigate the possible dose-dependent effects of mVNs on different physiological parameters in humans. 3 protocols of mVNs will be compared consisting of (1) 4 minutes (2 minutes on each side); (2) 12 minutes (3 sessions of 2 minutes of stimulation, with 2 minutes of rest for each side); (3) 16 minutes (8 minutes on each side). The following outcomes will be assessed before and after the stimulation: HR at rest, HRV, balance on standing, perceived intensity and modulation of mechanical stimuli on the skin of the forehead, and the abdomen, gastrointestinal transit, and a fecal sample from the closest intestinal emptying. A total sample of at least 96 healthy subjects (48 females) aged between 18 and 60 are expected to participate. The bidirectional communication between internal organs and the brain via the VN is a well-established scientific fact. Indeed, VNs has beneficial effects on manifold pathological conditions in humans. However, easy-to-apply, non-invasive, and effective VNs methods and standardized protocols are lacking. The here proposed project aims at refining and critically assessing mVNs methods - a prerequisite for exploring the clinical utility of mVNs and fostering its therapeutic potential given the fundamental role of the VN in regulating health and disease. Results obtained from this project will provide data on mVNs on gut microbiota dynamics and the potential benefits for pain modulation, equilibrium impairments, and gastrointestinal dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* agreement to participate by signing the informed consent form, being 18-60 years old, and sober

Exclusion Criteria:

* participants having significant neck pain, headache, or leg pain [with Numeric Pain Rating Scale (NPRS) greater than 3/10],
* pregnancy
* recent neck or cardiovascular surgery or significant trauma in the preceding 3 months
* diagnosis of cancer or inflammatory disorders (fever),
* spinal cord or cauda equina signs,
* widespread neurological disorders affecting the tone of the limbs and neck muscles
* underlying diseases, such as diabetes mellitus.
* pace-maker
* antibiotic prescription during the last 3 months
* gastrointestinal surgery,
* lower extremity injury (acute or overuse) that prevented them from participating in sports activities for at least one day in the previous 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate at rest | The outcome will be measured before the stimulation protocol and immediately after the stimulation protocol
  Heart rate is recorded continuously from 2 minutes before to 2 minutes after the stimulation using a fingertip infrared pulse oximeter. Heart rate will be measured in beats per minute.
Heart Rate Variability at rest | The outcome will be measured before the stimulation protocol and immediately after the stimulation protocol
  Polar H10 (1000 Hz) Chest Strap (rubber band placed comfortably around the chest above the xiphoid process level) for data acquisition will be worn by the participant for the duration of the assessment and the stimulation protocol. ECG waves will be acquired via Bluetooth to Elite HRV (Version 5.5.9, Asheville, NC, USA) on an Android device. HRV results from Elite HRV displayed on the app will be recorded for analysis with an Open HRV reading 2 minutes before the stimulation and 2 minutes immediately after. At the end of the data acquisition session, the chest strap will be removed. Distance between R peaks in the ECG, defined as RR Interval (Interbeat intervals [IBIs]) will be used as a reference to define HRV.
Mechanical Pain Intensity | The outcome will be measured before the stimulation protocol and immediately after the stimulation protocol
  These tests will be adopted to assess peripheral and central sensitization phenomena. Tests will be administered once for each site, using Neuropen with a Neurotip (disposable needle with a defined pressure of 40 g) and by applying 75 g pressure monofilament for 2 seconds on the skin site.
  If the stimulus is perceived as a pinprick by the participant, it will be requested to rate the pain intensity (NRS, "0 = no pain" to "10 = worst imaginable pain").

SECONDARY OUTCOMES:
Wind-up ratio | The outcome will be measured before the stimulation protocol and immediately after the stimulation protocol
  The temporal summation will be tested by comparing the pain rating of a single pinprick stimulus and a train of 10 pinprick stimuli of the same force repeated at a rate of 1/second using 75 g pressure monofilament on the same squared centimetre of skin area. The stimuli will be administered on the skin of the forehead (2 cm above the eyebrow and pupil center), on the neck above the middle of the sternocleidomastoideus muscle belly, and the abdomen (middle of the lines connecting the umbilicus to the anterior superior spina iliaca).
  If the stimulus is perceived as a pinprick by the participant, it will be requested to rate the pain intensity (NRS, "0 = no pain" to "10 = worst imaginable pain").
  The test will be repeated 5 times, and the mean pain rating of trains divided by a single stimulus was defined as the WUR.
One-leg support test | The outcome will be measured before the stimulation protocol and immediately after the stimulation protocol
  Balance will be tested by standing on the dominant leg with eyes closed, freeing the hands from a rail positioned in front of the participant, and maintaining the balance after the test has begun (hearing an acoustic signal). Further attempts can be performed until three successful attempts are completed without touching the ground with the non-dominant leg or opening the eyes for at least 20 seconds. During the test, participants are supported by an experimenter who stands next to them and is ready to provide assistance.
Mechanical pressure intensity | The outcome will be measured before the stimulation protocol and immediately after the stimulation protocol
  Participants' mechanical pressure intensity will be assessed by the intensity rate of the stimuli using a numerical rating scale (0-10 no pain - the worst ever imagined) on the skin of the forehead (2 cm above the eyebrow and pupil center), on the neck above the middle of the sternocleidomastoideus muscle belly, and the abdomen (middle of the lines connecting the umbilicus to the anterior superior spina iliaca) using a standardized pressure of 1 and 10 gr monofilament.
The Gastrointestinal Symptom Rating Scale | The outcome will be measured before the stimulation protocol, immediately after the stimulation protocol, and one week after the stimulation
  The scale consists of 13 items that assess the intensity of symptoms (each item is rated on a 7-point Likert scale; 1=No discomfort at all - 7= Very severe discomfort) related to gastrointestinal problems (i.e. possible symptoms such as difficulty or pain in digesting some foods; GSRS). The higher the score, the more gastrointestinal symptoms are present. A minimum score of 13 indicates no gastrointestinal symptoms. A maximum score of 101 indicates a severe presence of gastrointestinal symptoms.
The Bristol Stool Form Scale | The outcome will be measured for 1 week before and for 2 weeks after the administration of e week after the stimulation
  This validated scale allows determining whether digestion is normal, too slow or too fast based on the shape of the stool (BSFS). After a visual inspection of the stool, it is requested to give a rating using the shapes provided.
  The BSFS takes 30 seconds to complete and is required to complete the scale after the first bowel movement of the day. 7 type of stool are depicted and described. A sausage-shaped poop with cracks on the surface (Type 3) is considered normal on the Bristol Stool Scale. Type1-2 means too slow gastric transit while Type 4-7 too fast gastric transit.
  A sheet on which the daily scores will be reported by the participant will be provided after the agreement to participate and the signing of the informed consent.
Gut microbiota composition and function | The outcome will be measured before the stimulation protocol and immediately after the stimulation protocol
  Two stool sample kits will be provided to the participants so that they can collect a sample from the first bowel movement of the day and immediately after the stimulation protocol.
  Participants will be asked to bring the sample as soon as possible to the laboratory where they will be conserved and analysed. Metaproteomic analysis of each sample will be performed to estimate the gut microbiota composition by Shannon index to estimate the α-diversity (number of taxa/sample) and by Jaccard distance (defined as the ratio of taxa shared between samples/total number of taxa) to estimate the ß-diversity index. Gut microbiota function will be estimated by adopting the identified pathways of bacteria from the Kyoto Encyclopedia for Genes and Genomes (KEGG). The total protein intensity belonging to each pathway in each sample will be adopted for the analyses

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Carta, PhD, Principal Investigator — University of Vienna
Locations (1):
- UVienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. All of the individual participant data collected during the trial will be shared after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following the publication. No end date.
Access Criteria: The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.